CLINICAL TRIAL: NCT02172235
Title: Relative Bioavailability of Pioglitazone After Co-administration With Different Doses of BI 10773 in Healthy Volunteers (an Open-label, Randomised, Crossover, Clinical Phase I Study)
Brief Title: Relative Bioavailability of Pioglitazone After Co-administration With Different Doses of BI 10773 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1245.50
Record Dates: First submitted 2014-06-20; First posted 2014-06-24 (Estimated); Last update posted 2014-06-24 (Estimated); Status verified 2014-06

CONDITIONS: Healthy
MeSH Terms: interventions — Pioglitazone; empagliflozin

ARMS (6):
- Pioglitazone (Active Comparator)
  Interventions: Drug: Pioglitazone
- Pioglitazone + BI 10773 low (Experimental)
  Interventions: Drug: Pioglitazone; Drug: BI 10773 - low dose
- Pioglitazone + BI 10773 medium (Experimental)
  Interventions: Drug: Pioglitazone; Drug: BI 10773 - medium dose
- Pioglitazone + BI 10773 high (Experimental)
  Interventions: Drug: Pioglitazone; Drug: BI 10773 - high dose
- Pioglitazone low + BI 10773 medium (Experimental)
  Interventions: Drug: Pioglitazone - low dose; Drug: BI 10773 - medium dose
- Pioglitazone + BI 10773 1 hour after Pioglitazone (Experimental)
  Interventions: Drug: Pioglitazone; Drug: BI 10773 - medium dose

INTERVENTIONS:
Drug: Pioglitazone
  Arms: Pioglitazone; Pioglitazone + BI 10773 1 hour after Pioglitazone; Pioglitazone + BI 10773 high; Pioglitazone + BI 10773 low; Pioglitazone + BI 10773 medium
Drug: Pioglitazone - low dose
  Arms: Pioglitazone low + BI 10773 medium
Drug: BI 10773 - low dose
  Arms: Pioglitazone + BI 10773 low
Drug: BI 10773 - medium dose
  Arms: Pioglitazone + BI 10773 1 hour after Pioglitazone; Pioglitazone + BI 10773 medium; Pioglitazone low + BI 10773 medium
Drug: BI 10773 - high dose
  Arms: Pioglitazone + BI 10773 high

SUMMARY:
The objective was to investigate the effect of different doses of BI 10773 on the bioavailability of pioglitazone after multiple oral doses of both drugs

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male subjects according to the following criteria:

   medical history, physical examination, vital signs ((blood pressure (BP), pulse rate (PR), 12-lead electrocardiogram (ECG)), clinical laboratory tests
2. Age 18 to 55 years (incl.)
3. BMI 18.5 to 29.9 kg/m2 (incl.)
4. Signed and dated written informed consent prior to admission to the study in accordance with Good Clinical Practise (GCP) and the local legislation

Exclusion Criteria:

1. Any finding of the medical examination including blood pressure (BP), pulse rate (PR) and electrocardiogram (ECG) deviating from normal and of clinical relevance
2. Any evidence of a clinically relevant concomitant disease
3. Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
4. Surgery of the gastrointestinal tract (except appendectomy)
5. Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders
6. History of relevant orthostatic hypotension, fainting spells or blackouts.
7. Chronic or relevant acute infections
8. History of relevant allergy/hypersensitivity (including allergy to drug or its excipients)
9. Intake of drugs with a long half-life (more than 24 hours) within at least one month or less than 10 half-lives of the respective drug prior to administration or during the trial
10. Participation in another trial with an investigational drug within two months prior to administration or during the trial
11. Smoker (more than 10 cigarettes or more than 3 cigars or more than 3 pipes/day)
12. Inability to refrain from smoking on trial days
13. Alcohol abuse (more than 30 g/day)
14. Drug abuse
15. Blood donation (more than 100 mL within four weeks prior to administration or during the trial)
16. Excessive physical activities (within one week prior to administration or during the trial)
17. Alanine aminotransferase (ALT) outside the normal range or any other laboratory value outside the reference range that is of clinical relevance
18. Inability to comply with dietary regimen of trial site
19. Galactose or lactose intolerance, galactose or glucose malabsorption

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2010-04; Primary Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
AUCτ,ss (area under the concentration-time curve of the analyte in plasma at steady state over a uniform dosing interval τ) | Before each dosing, up to 10 days
Cmax,ss (maximum measured concentration of the analyte in plasma at steady state over a uniform dosing interval τ) | Before each dosing, up to 10 days

SECONDARY OUTCOMES:
C24,N (concentration of the analyte in plasma at 24 h after administration of the Nth dose) | Before each dosing, up to 10 days
λz (terminal elimination rate constant of the analyte in plasma) | Before each dosing, up to 10 days
t½ (terminal half-life of the analyte in plasma) | Before each dosing, up to 10 days
tmax (time from last dosing to maximum measured concentration of the analyte in plasma) | Before each dosing, up to 10 days
MRTpo (mean residence time of the analyte in the body at steady state after oral administration) | Before each dosing, up to 10 days
CL/F (apparent clearance of the analyte in the plasma after extravascular administration) | Before each dosing, up to 10 days
Vz/F (apparent volume of distribution during the terminal phase λz following extravascular administration) | Before each dosing, up to 10 days
Aet1-t2 (amount of analyte eliminated in urine over the time interval t1 to t2 ) | Day1 (-1-0, 0-4, 4-8, 8-12, and 12-24 h), Day 7 (143-144, 144-148, 148-152, 152-156, and 156-168 h)
fet1-t2 (fraction of dose excreted unchanged in urine over the time interval t1 to t2) | Day1 (-1-0, 0-4, 4-8, 8-12, and 12-24 h), Day 7 (143-144, 144-148, 148-152, 152-156, and 156-168 h)
CLR (renal clearance of the analyte in plasma afer extravascular administration) | Day1 (-1-0, 0-4, 4-8, 8-12, and 12-24 h), Day 7 (143-144, 144-148, 148-152, 152-156, and 156-168 h)
Cmax (maximum concentration of the analyte in plasma) | Before each dosing, up to 10 days
AUC0-tz (area under the concentration-time curve of the analyte in plasma over the time interval from 0 to the last quantifiable plasma concentration) | Before each dosing, up to 10 days
AUCτ,1 (area under the concentration-time curve of the analyte in plasma over the time interval from 0 to the last quantifiable plasma concentration within the first dosing interval) | Before each dosing, up to 10 days
AUC0-∞ (area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity) | Before each dosing, up to 10 days
Metabolite to parent ratio | Before each dosing, up to 10 days
Number of patients with abnormal findings in physical examination | up to 30 days after drug administration
Number of patients with abnormal changes in laboratory parameters | up to 30 days after drug administration
Number of patients with clinically significant changes in 12-lead electrocardiogram (ECG) | up to 30 days after drug administration
Number of patients with clinically significant changes in vital signs | up to 30 days after drug administration
Assessment of tolerability by investigator on a 4-point scale | up to 10 days
Number of patients with adverse events | up to 51 days